CLINICAL TRIAL: NCT00280878
Title: A Pilot Study of Rituximab in Combination With Out-patient Based VGF/F-GIV Salvage Therapies for Relapsed/Refractory CD20+ Lymphomas
Brief Title: Rituximab in Combination With Outpatient Therapy for CD20+ Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AH204/05
Record Dates: First submitted 2006-01-22; First posted 2006-01-24 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2007-10

CONDITIONS: Non-Hodgkin's Lymphoma (CD20+)
Keywords: Lymphoma; CD20+
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Gemcitabine; Vinorelbine; Ifosfamide; Rituximab

INTERVENTIONS:
Drug: gemcitabine
Drug: vinorelbine
Drug: ifosfamide
Drug: rituximab

SUMMARY:
This is a Phase II pilot study evaluating the safety of a risk-adjusted outpatient-based approach to lymphoma salvage therapy with VGF (vinorelbine, gemcitabine and pegfilgrastim) and/or F-GIV (gemcitabine, Ifosfamide, vinorelbine and pegfilgrastim) in combination with Rituximab (R-VGF/R-F-GIV).

DETAILED DESCRIPTION:
Recent epidemiologic surveys have demonstrated a dramatic increase in the incidence of non-Hodgkin's lymphoma (NHL). NHL is now one of the most rapidly increasing malignancies in the industrial world.

The purpose of this project is to evaluate the efficacy and safety of an outpatient treatment for relapsed or treatment resistant (refractory) CD20+ lymphoma. Two combinations of chemotherapy drugs will be tested depending on the patients prior therapy and response - rituximab, vinorelbine and gemcitabine (R-VGF) OR rituximab, vinorelbine, gemcitabine and ifosfamide (R-FGIV).

Previous experience, including a recently completed study using combinations of vinorelbine, gemcitabine and ifosfamide has demonstrated that such an outpatient approach is safe and of similar efficacy to presently available alternative inpatient chemotherapy approaches. This study is expanding on the findings from the previous study by adding rituximab.

Rituximab is being increasingly and successfully used in the therapy of CD20+ NHL. It is a specific protein (antibody) that is directed against the surface protein (CD20 antigen) found on CD20+ lymphoma cells and can therefore lead to the destruction of these cells. Rituximab also has a highly favourable toxicity profile enabling outpatient treatment.

All of these factors provide a strong rationale for the combination of rituximab and the novel outpatient-based salvage approaches VGF and F-GIV that we have recently evaluated. This pilot study of 12 patients will test the feasibility of this combination approach in patients with relapsed/refractory CD20+ NHL.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Relapsed or primary refractory CD20+ NHL
* ECOG 0 - 2
* Written informed consent

Exclusion Criteria:

* Intention to proceed with any form of transplant therapy following fewer than 2 cycles of protocol salvage therapy.
* Bilirubin > 50µmol/litre unless secondary to lymphoma
* Creatinine > 2 x upper limit of normal unless secondary to lymphoma
* Absolute neutrophil count <0.5 x 109/litre and / or platelets < 50 x 109/litre unless secondary to lymphoma
* Relapse within 6 months of a prior transplant procedure (autologous or allogeneic).
* Known sensitivity to E coli derived preparations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of a risk-adjusted outpatient-based approach to lymphoma salvage therapy with VGF and/or F-GIV in combination with Rituximab.

SECONDARY OUTCOMES:
To determine point estimates of the response rates achieved with R-VGF or R-F-GIV in previously treated patients with relapsed/refractory CD20+ B-cell NHL.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Spencer, Assoc.Prof, Study Chair
Locations (2):
- Australia (2):
  - The Alfred Hospital, Melbourne, Victoria
  - Frankston Hospital, Melbourne, Victoria